CLINICAL TRIAL: NCT03315091
Title: A Randomised, Open-label, Phase I Study to Determine the Effect of Food on the Pharmacokinetics of AZD1775 After Oral Dosing of a Capsule Formulation in Patients With Advanced Solid Tumours
Brief Title: Phase I Study to Assess the Effect of Food on AZD1775 Pharmacokinetics in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D6014C00005
Record Dates: First submitted 2017-09-28; First posted 2017-10-19 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Solid Tumours
Keywords: Pharmacokinetics, WEE1 inhibitor, food effect, safety assessments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment sequence 1 (Fasted-Fed) (Experimental): To assess the PK of AZD1775 following oral dosing of the capsule formulation in patients with advanced solid tumours in either a fed or fasted condition.
  Interventions: Drug: Treatment A - AZD1775 administered under fasted conditions; Drug: Treatment B - AZD1775 administered under fed conditions.
- Treatment sequence 2 (Fed-Fasted) (Experimental): To assess the PK of AZD1775 following oral dosing of the capsule formulation in patients with advanced solid tumours in either a fed or fasted condition.
  Interventions: Drug: Treatment A - AZD1775 administered under fasted conditions; Drug: Treatment B - AZD1775 administered under fed conditions.

INTERVENTIONS:
Drug: Treatment A - AZD1775 administered under fasted conditions — Premedication with Kytril (granisetron) 1 mg intravenously or Zofran (ondansetron) 8 mg intravenously within 30 to 40 minutes prior to administration of the AZD1775 capsules. Single dose 300 mg AZD1775, (3 x 100 mg, printed capsules) administered orally under fasted conditions. The drug class of AZD1775 is Wee-1 kinase inhibitor.
Drug: Treatment B - AZD1775 administered under fed conditions. — Premedication with Kytril (granisetron) 1 mg intravenously or Zofran (ondansetron) 8 mg intravenously within 30 to 40 minutes prior to administration of the AZD1775 capsules.
  Single dose 300 mg AZD1775, (3 x 100 mg, printed capsules) administered orally under fed conditions.
  The drug class of AZD1775 is Wee-1 kinase inhibitor.

SUMMARY:
The purpose of this study is to assess the effect of food on the pharmacokinetics (PK) of a single dose of AZD1775 (printed capsules) in patients with advanced solid tumours.

DETAILED DESCRIPTION:
This is a Phase I, open-label, randomised, 2-period crossover design study in patients with advanced solid tumours.

The purpose of this study is to assess the effect of food on the pharmacokinetics (PK) of a single dose of AZD1775 (printed capsules).In addition single dose safety and tolerability data will be gathered.

Patients will be screened within 28 days of Day 1 of the first treatment period (Period 1). Patients will take part in 2 randomised treatment sequences each separated by a washout period of at least 5 and no more than 14 days.

During Period 1, prior to administration of the first dose of study treatment, each patient will be randomised to 1 of 2 treatment sequences (Fasted-Fed or Fed-Fasted) to receive a single oral dose of 300 mg AZD1775 in each of the 2 treatment periods as follows:

* Fasted (Treatment A): Single dose 300 mg AZD1775, (3 x 100 mg, printed capsules).
* Fed (Treatment B): Single dose 300 mg AZD1775, (3 x 100 mg, printed capsules).

Pharmacokinetic and safety assessments will be obtained for up to 72 hours post-dose in each treatment period.

On completion of the study (ie, after collection of 72-hour PK sample and safety in period 2) patients will be evaluated per current assessments for their eligibility and interest to enrol into the open-label continued treatment access study (D6014C000007).

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study patients should fulfil the following criteria:

* Read and understand the informed consent form (ICF) and given written informed consent prior to any study procedures.
* Histologically or cytologically documented, locally advanced or metastatic solid tumour, excluding lymphoma, for which standard therapy does not exist or has proven ineffective or intolerable.
* Any prior palliative radiation must have been completed at least 7 days prior to the start of study treatment, and patients must have recovered from any acute adverse effects prior to the start of study treatment.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 to 1.
* Baseline laboratory values within 7 days of study treatment initiation:
* Absolute neutrophil count (ANC) ≥1500/μL.
* Haemoglobin ≥9 g/dL.
* Platelets ≥100,000/μL.
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 x upper limit of normal (ULN) or ≤5 x ULN if known hepatic metastases.
* Serum bilirubin within normal limits (WNL) or ≤1.5 x ULN in patients with liver metastases; or total bilirubin ≤3.0 x ULN with direct bilirubin WNL in patients with well documented Gilbert's Syndrome.
* Serum creatinine ≤1.5 x ULN, or measured creatinine clearance (CrCl) calculated by Cockcroft-Gault method ≥45 mL/min (confirmation of creatinine clearance is only required when creatinine is >1.5 x ULN) CrCl (glomerular filtration rate) = (140-age) x (weight/kg) x Fa (72 x serum creatinine mg/dL)

where F = 0.85 for females and F = 1 for males

* Female patients who are not of childbearing potential and fertile females of childbearing potential who agree to use adequate contraceptive measures that are in during screening (or consent), for the duration of the study, and for 1 month after treatment stops, and who are not breastfeeding, and who have a negative serum or urine pregnancy test prior to the start of study treatment.
* Male patients should be willing to use barrier contraception (ie, condoms) for the duration of the study and for 3 months after study treatment discontinuation
* Female or male patients ≥18 years.
* Patient should be able to adequately consume a high-fat meal as prescribed in Treatment B.
* Willingness and ability to comply with the study and the follow-up procedures.
* For inclusion in the optional genetic component of the study for all the patients:
* Provision of informed consent for genetic research. If a patient declines to participate in the genetic component of the study, there will be no penalty or loss of benefit to the patient. The patient will not be excluded from other aspects of the study described in the CSP, as long as all the eligibility criteria are met.

Exclusion Criteria:

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca personnel and/or personnel at the study centre).
* Previous enrolment or randomisation and received study treatment in the present study. Patients can, however, be re-screened if the reason for the screen failure no longer exists.
* Known malignant central nervous system (CNS) disease other than neurologically stable, treated brain metastases - defined as metastasis having no evidence of progression or haemorrhage for at least 2 weeks after treatment (including brain radiotherapy). Must be off any systemic corticosteroids for the treatment of brain metastases for at least 14 days prior to enrolment.
* Use of any anti-cancer treatment drug ≤21 days or 5 half-lives (whichever is shorter) prior to the first administration of AZD1775. For drugs for which 5 half lives is ≤21 days, a minimum of 10 days between termination of the prior treatment and administration of AZD1775 treatment is required.
* No other anticancer-therapy (chemotherapy, immunotherapy, hormonal anti-cancer therapy, radiotherapy [except for palliative local radiotherapy]), biological therapy or other novel agent is to be permitted while patient is receiving study treatment. Patients on LHRH analogue treatment for more than 6 months are allowed entry into the study and may continue at the discretion of the Investigator.
* Patients suffering from conditions which are likely to adversely affect gastrointestinal motility and/or transit (for example, diarrhoea, vomiting or nausea, gastroparesis, irritable bowel syndrome and malabsorption) or patients with gastrointestinal resection (eg, partial or total gastrectomy) likely to interfere with absorption of study treatment.
* Major surgical procedures ≤28 days of beginning study treatment, or minor surgical procedures ≤7 days. No waiting period required following port-a-cath placement or other central venous access placement.
* Grade >1 toxicities from prior therapy, according to the Common Terminology Criteria for Adverse Events (CTCAE), excluding alopecia or anorexia.
* Patient has an inability to swallow oral medications. Note: Patient may not have a percutaneous endoscopic gastrostomy tube or be receiving total parenteral nutrition.
* Patients who are not non-smokers or light smokers (no more than 5 cigarettes per day) and who cannot abstain from smoking from 2 weeks prior to the first administration of AZD1775 until after the last PK sample collection in Period 2.
* Any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of the first administration of AZD1775.
* Patient has had prescription or non-prescription drugs or other products known to be sensitive to cytochrome P450 (CYP)3A4 substrates or CYP3A4 substrates with a narrow therapeutic index, or to be moderate to strong inhibitors/inducers of CYP3A4 which cannot be discontinued 2 weeks prior to Day 1 of dosing and withheld throughout the study until 2 weeks after the last administration of AZD1775. Co administration of aprepitant or fosaprepitant during this study is prohibited
* Patient has had adjustments to prescription or non-prescription drugs or other products known to be weak inhibitors and/or inducers of CYP3A4 within 1 week prior to the first administration of AZD1775.
* Herbal preparations taken within 7 days of study entry. However, in the case of St John's wort, patients cannot have taken this herbal preparation 21 days prior to first administration of AZD1775.
* Patients who have taken any proton pump inhibitors (omeprazole, lansoprazole, esomeprazole, pantoprazole, etc) within 7 days of first administration of AZD1775.
* Patients who are dependent on a medication which could adversely affect gastrointestinal motility or transit (for example: diphenoxylate, [loperamide], metoclopramide, cisapride, tegaserod, erythromycin). Note that use of loperamide is permitted during the study for treatment of diarrhoea Narcotics that are not in the list of prohibited medications are allowed.
* Patients who cannot withhold antacids for 6 hours or H2-antagonists (cimetidine, ranitidine, famotidine, nizatidine) for 48 hours.
* Patients unable to fast for up to 14 hours.
* Patients with type 1 diabetes mellitus.
* Any known hypersensitivity or contraindication to AZD1775 or to the components thereof.
* Any of the following cardiac diseases currently or within the last 6 months as defined by the New York Heart Association ≥ Class 2.
* Unstable angina pectoris.
* Congestive heart failure.
* Acute myocardial infarction.
* Conduction abnormality not controlled with pacemaker or medication.
* Significant ventricular or supraventricular arrhythmias (patients with chronic rate controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible).
* AZD1775 should not be given to patients who have a history of Torsades de pointes unless all risk factors that contributed to Torsades have been corrected. AZD1775 has not been studied in patients with ventricular arrhythmias or recent myocardial infarction.
* Patients with QT interval (specifically QTc calculated using the Fridericia formula [QTcF] >450 ms/male and >470 ms/female) obtained from 3 electrocardiograms (ECGs) 2 to 5 minutes apart at study entry, or congenital long QT syndrome.
* Pregnant or lactating female patients.
* Serious, symptomatic active infection at the time of study entry, or another serious underlying medical condition that would impair the ability of the patient to receive study treatment.
* Active infection with hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).
* Any of the following is regarded as a criterion for exclusion from the optional pharmacogenetic part of the study:
* Previous bone marrow transplant.
* Non-leukocyte depleted blood product within 120 days of the genetic sample collection.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from zero to infinity for AZD1775 | Blood samples are collected on Day 1 of each treatment period at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours post AZD1775 dose
  To investigate the effect of food on the PK of a single dose of AZD1775 printed capsules following oral dosing in patients with advanced solid tumours
Area under the plasma concentration-time curve from time zero to the time "t" (AUC0-t) of the last quantifiable concentration for AZD1775 | Blood samples are collected on Day 1 of each treatment period at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours post AZD1775 dose
  To investigate the effect of food on the PK of a single dose of AZD1775 printed capsules following oral dosing in patients with advanced solid tumours
Cmax: maximum plasma drug concentration for AZD1775 | Blood samples are collected on Day 1 of each treatment period at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours post AZD1775 dose
  To investigate the effect of food on the PK of a single dose of AZD1775 printed capsules following oral dosing in patients with advanced solid tumours

SECONDARY OUTCOMES:
tmax,: time to reach maximum plasma concentration for AZD1775 | Blood samples are collected on Day 1 of each treatment period at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours post AZD1775 dose
  To characterise the PK of a single dose of AZD1775 printed capsules following oral dosing in patients with advanced solid tumours
λz: Elimination rate constant for AZD1775 | Blood samples are collected on Day 1 of each treatment period at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours post AZD1775 dose
  To characterise the PK of a single dose of AZD1775 printed capsules following oral dosing in patients with advanced solid tumours
Apparent clearance following oral administration for AZD1775 | Blood samples are collected on Day 1 of each treatment period at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours post AZD1775 dose
  To characterise the PK of a single dose of AZD1775 printed capsules following oral dosing in patients with advanced solid tumours
t½,: terminal half-life for AZD1775 | Blood samples are collected on Day 1 of each treatment period at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours post AZD1775 dose
  To characterise the PK of a single dose of AZD1775 printed capsules following oral dosing in patients with advanced solid tumours
Apparent volume of distribution for AZD1775 | Blood samples are collected on Day 1 of each treatment period at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours post AZD1775 dose
  To characterise the PK of a single dose of AZD1775 printed capsules following oral dosing in patients with advanced solid tumours
Adverse Events, graded by the National Cancer Institute Common Terminology Criteria for Adverse Event's (CTCAE v4.3) | Until 30 days following the final dose of AZD1775
  To assess the safety and tolerability of a single dose of AZD1775 printed capsules following oral dosing in patients with advanced solid tumours.
Complete physical examination including performance status assessed using the Eastern Cooperative Oncology Group (ECOG) Performance Status criteria. | Until 30 days following the final dose of AZD1775
  To assess the safety and tolerability of a single dose of AZD1775 printed capsules following oral dosing in patients with advanced solid tumours. If new or aggravated physical findings imply deterioration compared with baseline, the finding will be reported as an Adverse Event.
Pulse Rate (beats/min) | Until 30 days following the final dose of AZD1775
  To assess the safety and tolerability of a single dose of AZD1775 printed capsules following oral dosing in patients with advanced solid tumours.
Evaluation of Haematology Parameters (Haemoglobin, Leukocyte and Leukocyte counts, Red blood cell count, Haematocrit and Platelet Count) | Until 30 days following the final dose of AZD1775
  Laboratory tests will be performed by an accredited laboratory. Deterioration of haematology laboratory values as compared to baseline will be reported as Adverse Events if they fulfill any of the Serious Adverse Events criteria or are the reason for discontinuation of the study treatment unless clearly due to the progression of disease under study. If deterioration in a laboratory value is associated with clinical signs and symptoms, the sign or symptom will be reported as an AE and the associated laboratory result will be considered as additional information.
Electrocardiogram (ECG) - A 12-lead safety ECG (paper ECG printout of 10 seconds for Investigator review) | Until 7 days following the final dose of AZD1775
  To assess the safety and tolerability of a single dose of AZD1775 printed capsules following oral dosing in patients with advanced solid tumours. The Investigator will judge the overall interpretation as normal or abnormal. If abnormal, it will be decided as to whether or not the abnormality is clinically significant or not clinically significant.
Blood Pressure (mm Hg) | Until 30 days following the final dose of AZD1775
  To assess the safety and tolerability of a single dose of AZD1775 printed capsules following oral dosing in patients with advanced solid tumours.
Body Temperature (°C) | Until 30 days following the final dose of AZD1775
  To assess the safety and tolerability of a single dose of AZD1775 printed capsules following oral dosing in patients with advanced solid tumours.
Evaluation of Clinical Chemistry Parameters (Albumin, Alanine Transaminase, Aspartate Transaminase, Alkaline Phosphatase, Bilirubin, Calcium, Creatinine, Glucose, Total protein, Chloride, Potassium, Sodium, Urea nitrogen) | Until 30 days following the final dose of AZD1775
  Laboratory tests will be performed by an accredited laboratory. Deterioration of clinical chemistry values as compared to baseline will be reported as Adverse Events if they fulfil any of the Serious Adverse Events criteria or are the reason for discontinuation of the study treatment unless clearly due to the progression of disease under study.
  If deterioration in a laboratory value is associated with clinical signs and symptoms, the sign or symptom will be reported as an AE and the associated laboratory result will be considered as additional information.

CONTACTS AND LOCATIONS:
Overall Officials: Lone Ottesen, MD, Study Director — AstraZeneca; Henk Verheul, MD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (6):
- France (2):
  - Research Site, Bordeaux
  - Research Site, Saint-Herblain
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Maastricht
- United Kingdom (2):
  - Research Site, Glasgow
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: No